CLINICAL TRIAL: NCT03714672
Title: A Randomized, Double-blind, Multi-site, Comparator-controlled, Phase III Trial to Evaluate the Efficacy and Safety of a Fixed-dose Combination of Tramadol Hydrochloride and Diclofenac Sodium in Acute Moderate to Severe Pain After Third Molar Extraction
Brief Title: Tramadol/Diclofenac Fixed-dose Combination Phase III Trial in Acute Pain After Third Molar Extraction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Collaborators: Grünenthal, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KF8001-01; U1111-1179-2333 (Other: World Health Organization); KF8001-01 (Registry Identifier: RNEC (Mexico))
Record Dates: First submitted 2018-10-19; First posted 2018-10-22 (Actual); Results first posted 2019-07-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Acute Pain
Keywords: Wisdom tooth removal; Dental pain
MeSH Terms: conditions — Acute Pain; Toothache | interventions — Tramadol; Diclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study used double-blind and double-dummy methods to guarantee the blinding of all personnel involved in the study. Participants, investigators, and all persons involved in the conduct, data management, and analysis of the study were fully blinded to the participant's treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Tramadol/Diclofenac 50/50 (Experimental): Participants received 3 doses of tramadol hydrochloride/diclofenac sodium 50 mg/50 mg over a 24-hour period if they developed acute moderate to severe pain within 4 hours after third molar extraction.
  Interventions: Drug: Tramadol/Diclofenac 50/50
- Tramadol/Diclofenac 25/25 (Experimental): Participants received 3 doses of tramadol hydrochloride/diclofenac sodium 25 mg/25 mg over a 24-hour period if they developed acute moderate to severe pain within 4 hours after third molar extraction.
  Interventions: Drug: Tramadol/Diclofenac 25/25
- Tramadol 50 (Active Comparator): Participants received 3 doses of tramadol hydrochloride 50 mg over a 24-hour period if they developed acute moderate to severe pain within 4 hours after third molar extraction.
  Interventions: Drug: Tramadol 50
- Diclofenac 50 (Active Comparator): Participants received 3 doses of diclofenac sodium 50 mg over a 24-hour period if they developed acute moderate to severe pain within 4 hours after third molar extraction
  Interventions: Drug: Diclofenac 50

INTERVENTIONS:
Drug: Tramadol/Diclofenac 50/50 — Each dose comprised 1 fixed-dose combination tablet and 3 placebo tablets or capsules matching the other active treatment groups. Doses were taken 8 hours apart.
  Other Names: Adorlan Forte (Registered Trademark)
  Arms: Tramadol/Diclofenac 50/50
Drug: Tramadol/Diclofenac 25/25 — Each dose comprised 1 fixed-dose combination tablet and 3 placebo tablets or capsules matching the other active treatment groups. Doses were taken 8 hours apart.
  Other Names: Adorlan (Registered Trademark)
  Arms: Tramadol/Diclofenac 25/25
Drug: Tramadol 50 — Each dose comprised 1 capsule containing 50 mg tramadol hydrochloride and 3 placebo tablets matching the other active treatment groups. Doses were taken 8 hours apart.
  Other Names: Tramadol immediate-release capsule; Tradol (Registered Trademark)
  Arms: Tramadol 50
Drug: Diclofenac 50 — Each dose comprised 1 tablet containing 50 mg diclofenac sodium and 3 placebo tablets or capsules matching the other active treatment groups. Doses were taken 8 hours apart.
  Other Names: Voltaren (Registered Trademark) (diclofenac enteric-coated tablet)
  Arms: Diclofenac 50

SUMMARY:
This study evaluated a new drug fixed-dose combination tablet (FDC) called tramadol/diclofenac at two different strengths (fixed doses of 25 milligrams [mg] of tramadol and of diclofenac or of 50 mg each). Tramadol and diclofenac each relieve pain, but they do so by different mechanisms. They were used alone as comparator drug in this study. Both are marketed drugs and are standard treatment for acute pain, including wisdom tooth removal.

DETAILED DESCRIPTION:
The purpose of this study was to demonstrate that the FDC of Tramadol and Diclofenac 50/50 has superior analgesic effect than the monotherapies and that the FDC of Tramadol and Diclofenac 25/25 has non-inferior analgesic effect than the monotherapies. There was an Enrollment Period, a blinded Treatment Period, and a Follow-up Period. Previously used analgesic medication was washed out for at least 24 hours before surgery. The Treatment Period starts on Day 1 with dental surgery and treatment allocation. Treatment was started within 4 hours after the end of surgery if the participant's pain intensity had reached at least 5 points on the 11-point numerical rating scale (NRS). Each participant received 3 doses of one of the four treatments within 24 hours. One fourth of the participants received the fixed-dose combination tablet at a low dose, one fourth at the higher dose, one fourth received 50 mg of the comparator tramadol alone, and one fourth 50 mg of the comparator diclofenac alone.

The first 2 doses of the investigational medicinal product (IMP) were taken at the site, the last dose in an out-patient setting. Participants returned to the site at 24 hours after the first dose. A Follow-up Period included a final visit at the site or a phone call on Day 14 to assess the participant's safety.

ELIGIBILITY:
Inclusion Criteria:

1. The participant has read the informed consent form, has understood the relevant aspects of the clinical study, and grants his/her authorization to participate by signing the informed consent form prior to the inclusion in the clinical study and the performance of any procedure.
2. Male and female participants above 18 years up to 60 years.
3. Female participants of childbearing potential must be practicing an acceptable method of birth control and must have a negative urine pregnancy test at enrollment with confirmation at the Allocation Visit.
4. Participants are in good health, i.e., the medical record, vital signs, physical examination, and laboratory parameter assessments do not show any abnormal deviations impeding the participation in the clinical study.
5. Participants requiring extraction of 3 or more third molars with 2 mandibular impacted third molars.
6. Clinical and radiological diagnosis of impacted lower third molars.
7. Class I and Class II molars according to Pell and Gregory's classification (Gay Escoda et al. 2004).
8. Participants must be able to swallow the IMPs.

Exclusion Criteria at Enrollment:

1. Findings in the medical record, vital signs, and/or physical examination demonstrating abnormal conditions of participant's general state of health preventing his/her participation in the clinical study according to the investigator's opinion.
2. Participant unable to speak, read, or write in Spanish language.
3. Clinical laboratory parameters exceed the pre-defined alert ranges (i.e., 1 standard deviation above or below the upper/lower limit of the normal ranges).
4. Known hypersensitivity to the IMPs, the anesthetic to be used during surgery, or to the rescue medication (ibuprofen, ketorolac).
5. Known alcohol or drug abuse in the last 6 months or any history of seizures. Alcohol abuse is defined as the consumption of more than 3 ounces (about 90 milliliters) of liquor or spirits or 18 ounces (about 530 milliliters) of beer per day, for 5 consecutive days during the 6-month period. Drug abuse is defined as the use of any recreational drug for 5 consecutive days during the 6 month period.
6. Participants who take analgesic medication for chronic pain, monoamine oxidase inhibitors, tricyclic antidepressants, neuroleptics, or other drugs that reduce the seizure threshold within 4 weeks of enrollment.
7. Pregnant or lactating women.
8. Participants who received systemic corticosteroids or opioid analgesics less than 2 weeks before surgery.
9. Participants with molars linked to the mandibular canal.
10. Participants requiring immediate dental procedures other than third and fourth molars extraction,

    Exclusion Criteria at the Allocation Visit:
11. Participant received a long-acting non-steroidal anti-inflammatory drug within 24 hours or 5 times the elimination half-life of that drug prior to surgery, whatever the longer.
12. Participant received any analgesic medication other than short-acting pre-operative or intra-operative anesthetic agents within 24 hours before taking IMPs.
13. Participant received more than 300 mg of lidocaine in total.
14. Participant received any analgesic medication other than the IMPs immediately after the oral surgical procedure was completed.
15. Baseline pain intensity of the participant after oral surgical procedure remains below 5 points on the 11-point NRS.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1151 (Actual)
Dates: Start 2017-08-26 (Actual); Primary Completion 2018-03-09 (Actual); Study Completion 2018-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grünenthal Study Director, Study Director — Grünenthal GmbH
Locations (7):
- Mexico (7):
  - Private Clinic, Zapopan, Jalisco
  - Private Clinic, Monterrey, Nuevo León
  - Private Clinic, Aguascalientes
  - Private Clinic, Chihuahua City
  - Private Clinic, León
  - Private Clinic, Puebla City
  - University, San Luis Potosí City

IPD SHARING:
Plan to Share IPD: Yes
Information available on the Grünenthal Group Web Site (see URL below for details).
Supporting Information: Study Protocol, SAP, CSR
URL: http://www.grunenthal.com/r-d-vision-mission/clinical-trials/data-sharing-clinical-trials

REFERENCES:
- [Background] Gay Escoda C, Piñera Penalva M, Velasco Vivancos V, Berini Aytés L. Cordales incluidos. Patología, clínica y tratamiento del tercer molar incluído. In: Gay Escoda C, Berini Aytés L. (eds.). Tratado de Cirugía Bucal. Tomo I. Madrid: Ergón; 2004. p. 355-85

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant was enrolled on 26 August 2017.
Pre-assignment Details: A total of 1151 participants signed an informed consent form, 829 participants were allocated to treatment. Of the 829 allocated participants, 3 were not treated (1 each in the Diclofenac 50, Tramadol 50, and Tramadol/Diclofenac 25/25 treatment arms) and were not included in the Safety Set (N=826).
Period: Overall Study
Arm/Group | Tramadol/Diclofenac 50/50 | Tramadol/Diclofenac 25/25 | Tramadol 50 | Diclofenac 50
Started | 209 | 206 | 206 | 208
Safety Set | 208 | 205 | 206 | 207
Completed | 207 | 202 | 202 | 207
Not Completed | 2 | 4 | 4 | 1
Not completed — Adverse Event | 0 | 0 | 3 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Other Reason | 1 | 2 | 1 | 1
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Set (One participant was allocated to Tramadol/Diclofenac 50/50, but received Tramadol 50. The participant was included in the Tramadol 50 arm for the Safety Set as the analyses were conducted according to the treatment received)
Groups:
- Tramadol 50: Participants received 3 doses of tramadol hydrochloride 50 mg over a 24-hour period if they developed acute moderate to severe pain within 4 hours after third molar extraction.
  Tramadol 50: Each dose comprised 1 capsule containing 50 mg tramadol hydrochloride and 3 placebo tablets matching the other active treatment groups. Doses were be taken 8 hours apart.
- Diclofenac 50: Participants received 3 doses of diclofenac sodium 50 mg over a 24-hour period if they developed acute moderate to severe pain within 4 hours after third molar extraction
  Diclofenac 50: Each dose comprised 1 tablet containing 50 mg diclofenac sodium and 3 placebo tablets or capsules matching the other active treatment groups. Doses were be taken 8 hours apart.
- Total: Total of all reporting groups
Arm/Group | Tramadol/Diclofenac 50/50 | Tramadol/Diclofenac 25/25 | Tramadol 50 | Diclofenac 50 | Total
Number analyzed (Participants) | 208 | 205 | 206 | 207 | 826
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 208 | 205 | 206 | 207 | 826
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 22.9 [18 to 41] | 24.0 [18 to 50] | 23.8 [18 to 41] | 23.6 [18 to 56] | 23.6 [18 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 136 | 132 | 135 | 529
  Male | 82 | 69 | 74 | 72 | 297
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 208 | 204 | 206 | 206 | 824
  Not Hispanic or Latino | 0 | 1 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 0 | 1 | 3
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 4 | 4 | 2 | 10
  More than one race | 202 | 198 | 200 | 203 | 803
  Unknown or Not Reported | 6 | 1 | 2 | 1 | 10
Region of Enrollment [Number; unit: participants]
  Mexico | 208 | 205 | 206 | 207 | 826
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.5 (4.08) | 25.0 (4.39) | 25.1 (4.25) | 24.5 (4.51) | 24.8 (4.31)
Baseline pain intensity categorized [Count of Participants; unit: Participants] — Measured using an 11-point NRS by answering the following question: "Please rate your pain by selecting the one number that best describes how much pain you have right now." Scores ranged from 0 (no pain) to 10 (pain as bad as you can imagine, and were categorized as None (0), Mild (≥ 1 and < 5), Moderate (≥ 5 and ≤ 6), and Severe (≥ 7). Baseline was the score assessed before the first dose of IMP.
  Participants
    Moderate | 88 | 87 | 86 | 81 | 342
    Severe | 120 | 117 | 120 | 126 | 483
    None | 0 | 0 | 0 | 0 | 0
    Mild | 0 | 0 | 0 | 0 | 0
    Missing | 0 | 1 | 0 | 0 | 1
Baseline pain intensity 11-point NRS [Mean (Standard Deviation); unit: units on a scale] — Measured using an 11-point NRS by answering the following question: "Please rate your pain by selecting the one number that best describes how much pain you have right now." Scores ranged from 0 (no pain) to 10 (pain as bad as you can imagine, and were categorized as None (0), Mild (≥ 1 and < 5), Moderate (≥ 5 and ≤ 6), and Severe (≥ 7). Baseline was the score assessed before the first dose of IMP. Population: One participant (Tramadol/Diclofenac 25/25) from the Safety Set had no efficacy assessments and was not included in the Full Analysis Set.
  units on a scale
    number analyzed (Participants) | 208 | 204 | 206 | 207 | 825
    (all) | 7.0 (1.51) | 7.0 (1.45) | 7.0 (1.45) | 7.0 (1.40) | 7.0 (1.45)
Number of molars extracted [Count of Participants; unit: Participants]
  Number of molars extracted 3 | 37 | 41 | 42 | 43 | 163
  Number of molars extracted 4 | 171 | 164 | 164 | 164 | 663
Duration of surgery, minutes [Mean (Standard Deviation); unit: minutes] | 33.0 (21.90) | 35.0 (21.56) | 34.2 (20.25) | 32.9 (19.21) | 33.8 (20.74)
Lidocaine used during surgery, mg [Mean (Standard Deviation); unit: mg] | 211.1 (44.18) | 211.4 (41.13) | 211.3 (43.36) | 207.7 (42.13) | 210.4 (42.67)
End of surgery to first dose of IMP, hours [Mean (Standard Deviation); unit: hours] | 2.2 (0.89) | 2.2 (0.83) | 2.1 (0.90) | 2.1 (0.85) | 2.2 (0.87)

OUTCOME MEASURES:

1. Primary Outcome: Pain Relief Expressed as Total Pain Relief (TOTPAR) Over the 4 Hours Post-dose Period (TOTPAR4)
Description: Pain relief was assessed by the participant at defined time points after the first IMP dose using a 5-point verbal rating scale (VRS) with categories 0 (none), 1 (a little), 2 (some), 3 (a lot), or 4 (complete). Total Pain Relief (TOTPAR4) is a time-weighted summary measure of the total area under the pain relief curve that integrates serial assessments of a participant's pain over the duration of 4 hours after IMP intake. Minimum and maximum values for TOTPAR4 were 0=worst score and 16=best score, a higher score indicates more pain relief.
Time Frame: Up to 4 hours after first dose
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tramadol/Diclofenac 50/50 | Tramadol/Diclofenac 25/25 | Tramadol 50 | Diclofenac 50
Number analyzed (Participants) | 209 | 204 | 205 | 207
units on a scale | 9.9 [9.3 to 10.4] | 8.6 [8.0 to 9.1] | 5.4 [4.9 to 5.9] | 5.8 [5.3 to 6.3]
Statistical Analysis 1: Comparison: Tramadol/Diclofenac 50/50 vs Diclofenac 50; Bonferroni-Holm procedure used for determining the statistical significance of the results; Test type: Superiority; p < 0.0001, ANCOVA; ANCOVA model with treatment, baseline pain intensity, and site as covariates; Mean Difference (Final Values) = -4.1, 95% CI 2-sided [-4.8 to -3.4] — LS means, 95% CIs, and pairwise CIs and p-values comparing the combination treatment arm to the monotherapy arm
Statistical Analysis 2: Comparison: Tramadol/Diclofenac 50/50 vs Tramadol 50; Bonferroni-Holm procedure used for determining the statistical significance of the results; Test type: Superiority; p < 0.0001, ANCOVA; ANCOVA model with treatment, baseline pain intensity, and site as covariates; Mean Difference (Final Values) = -4.5, 95% CI 2-sided [-5.2 to -3.8] — LS means, 95% CIs, and pairwise CIs and p-values comparing the combination treatment arm to the monotherapy arm
Statistical Analysis 3: Comparison: Tramadol/Diclofenac 25/25 vs Tramadol 50; Bonferroni-Holm procedure used for determining the statistical significance of the results. The planned test was a test for non-inferiority; Test type: Superiority; p < 0.0001, ANCOVA; ANCOVA model with treatment, baseline pain intensity, and site as covariates; Mean Difference (Final Values) = -3.2, 95% CI 2-sided [-3.9 to -2.5] — LS means, 95% CIs, and pairwise CIs and p-values comparing the combination treatment arm to the monotherapy arm
Statistical Analysis 4: Comparison: Tramadol/Diclofenac 25/25 vs Diclofenac 50; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p < 0.0001, ANCOVA; ANCOVA model with treatment, baseline pain intensity, and site as covariates; Mean Difference (Final Values) = -2.8, 95% CI 2-sided [-3.5 to -2.1] — LS means, 95% CIs, and pairwise CIs and p-values comparing the combination treatment arm to the monotherapy arm

2. Secondary Outcome: Total Pain Relief at 6 Hours Post-dose (TOTPAR6)
Description: Pain relief was assessed by the participant at defined time points after the first IMP dose using a 5-point VRS with categories 0 (none), 1 (a little), 2 (some), 3 (a lot), or 4 (complete). Total Pain Relief (TOTPAR6) is a time-weighted summary measure of the total area under the pain relief curve that integrates serial assessments of a participant's pain over the duration of 6 hours after IMP intake. Minimum and maximum values for TOTPAR6 were 0=worst score and 24=best score, a higher score indicates more pain relief.
Time Frame: Up to 6 hours after first dose
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tramadol/Diclofenac 50/50 | Tramadol/Diclofenac 25/25 | Tramadol 50 | Diclofenac 50
Number analyzed (Participants) | 209 | 204 | 205 | 207
units on a scale | 15.2 [14.4 to 16.0] | 13.3 [12.5 to 14.2] | 9.3 [8.4 to 10.1] | 9.8 [9.0 to 10.6]

3. Secondary Outcome: Total Pain Relief at 8 Hours Post-dose (TOTPAR8)
Description: Pain relief was assessed by the participant at defined time points after the first IMP dose using a 5-point VRS with categories 0 (none), 1 (a little), 2 (some), 3 (a lot), or 4 (complete). Total Pain Relief (TOTPAR8) is a time-weighted summary measure of the total area under the pain relief curve that integrates serial assessments of a participant's pain over the duration of 8 hours after IMP intake. Minimum and maximum values for TOTPAR8 were 0=worst score and 32=best score, a higher score indicates more pain relief.
Time Frame: Up to 8 hours after first dose
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tramadol/Diclofenac 50/50 | Tramadol/Diclofenac 25/25 | Tramadol 50 | Diclofenac 50
Number analyzed (Participants) | 209 | 204 | 205 | 207
units on a scale | 20.1 [19.0 to 21.2] | 17.8 [16.7 to 18.9] | 13.1 [12.0 to 14.2] | 13.7 [12.6 to 14.8]

4. Secondary Outcome: Summed Pain Intensity Difference (SPID) at 4, 6, 8, and 24 Hours Post-dose
Description: Pain intensity was assessed by the participant before and at defined time points after the first IMP dose using an 11-point NRS with anchors at 0 for "no pain" and 10 for "pain as bad as you can imagine". Pain Intensity Difference (PIDt) was defined as the difference between baseline pain intensity and pain intensity at time point t, and SPID defined as summed PIDt x [time (hours) elapsed since previous observation]. The SPID scores are the sum of the differences at each time point multiplied by the duration in hours since the previous time point. Positive numbers indicate a reduction in pain [maximum=10 at each time point], and negative numbers indicate an increase in pain [minimum=-10 at each time point]. The overall minimum and maximum are -10 and 10 times the number of hours specified (SPID-4=[-40 to 40], SPID-6=[-60 to 60], SPID-8=[-80 to 80], and SPID-24=[-240 to 240]).
Time Frame: Baseline; up to 24 hours after first dose
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tramadol/Diclofenac 50/50 | Tramadol/Diclofenac 25/25 | Tramadol 50 | Diclofenac 50
Number analyzed (Participants) | 209 | 204 | 205 | 207
units on a scale
  4 Hours | 16.24 (0.564) | 13.67 (0.576) | 6.43 (0.570) | 7.72 (0.568)
  6 Hours | 25.54 (0.836) | 21.86 (0.855) | 12.89 (0.845) | 14.36 (0.843)
  8 Hours | 33.70 (1.121) | 28.90 (1.146) | 19.10 (1.133) | 20.54 (1.129)
  24 Hours | 107.15 (3.787) | 91.99 (3.873) | 71.41 (3.828) | 72.08 (3.816)

5. Secondary Outcome: Time to Achieve a 50 Percent Reduction in Baseline Pain (Pain at Least Half Gone)
Description: Time (hours) when the participant achieved a 50 percent reduction of baseline (starting) pain. It was assessed at defined time points after the first IMP dose using a YES or NO question for pain half gone.
Time Frame: Up to 24 hours after first dose
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Tramadol/Diclofenac 50/50 | Tramadol/Diclofenac 25/25 | Tramadol 50 | Diclofenac 50
Number analyzed (Participants) | 209 | 204 | 205 | 207
hours | 1.27 (1.216) | 1.73 (2.778) | 3.01 (3.731) | 2.53 (2.865)

6. Secondary Outcome: Time to Onset of First Perceptible Pain Relief
Description: Participants used one stopwatch to document the time between first IMP dose and when they begin to feel any pain-relieving effect from the IMP.
Time Frame: Up to 8 hours after first dose
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Tramadol/Diclofenac 50/50 | Tramadol/Diclofenac 25/25 | Tramadol 50 | Diclofenac 50
Number analyzed (Participants) | 209 | 204 | 205 | 207
hours | 0.57 (0.483) | 0.67 (0.875) | 1.07 (1.000) | 1.12 (1.151)

7. Secondary Outcome: Time to Onset of Meaningful Pain Relief
Description: Participants used a second stopwatch to document the time between first IMP dose and when they felt their pain relief was meaningful to them.
Time Frame: Up to 8 hours after first dose
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Tramadol/Diclofenac 50/50 | Tramadol/Diclofenac 25/25 | Tramadol 50 | Diclofenac 50
Number analyzed (Participants) | 209 | 204 | 205 | 207
hours | 1.47 (1.149) | 2.04 (1.810) | 2.93 (1.895) | 2.75 (1.882)

8. Secondary Outcome: Time to Intake of First Rescue Medication Dose
Description: The time from first IMP dose to first dose of rescue medication (ibuprofen or ketorolac), if needed, within 24 hours post-dose was calculated.
Time Frame: First dose to 24 hours after first dose
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Tramadol/Diclofenac 50/50 | Tramadol/Diclofenac 25/25 | Tramadol 50 | Diclofenac 50
Number analyzed (Participants) | 209 | 204 | 205 | 207
hours | 21.84 (6.222) | 20.99 (7.450) | 17.37 (9.745) | 17.38 (9.646)

9. Secondary Outcome: Subject's Global Evaluation of the Treatment
Description: Participants documented their overall impression of the analgesic efficacy of the IMPs on a 5-point Likert scale from Excellent (4) to Poor (0).
Time Frame: 8 hours after the first dose of IMP or before first intake of rescue medication (whatever the first) and 24 hours after the first dose of IMPs
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Tramadol/Diclofenac 50/50 | Tramadol/Diclofenac 25/25 | Tramadol 50 | Diclofenac 50
Number analyzed (Participants) | 209 | 204 | 205 | 207
Participants
  8-Hours: number analyzed (Participants) | 207 | 199 | 197 | 201
  8-Hours: Poor | 4 | 7 | 28 | 23
  8-Hours: Fair | 10 | 12 | 30 | 25
  8-Hours: Good | 17 | 33 | 36 | 35
  8-Hours: Very Good | 73 | 64 | 52 | 67
  8-Hours: Excellent | 103 | 83 | 51 | 51
  24-Hours: number analyzed (Participants) | 208 | 201 | 205 | 206
  24-Hours: Poor | 3 | 4 | 7 | 7
  24-Hours: Fair | 4 | 5 | 23 | 13
  24-Hours: Good | 12 | 18 | 34 | 39
  24-Hours: Very Good | 57 | 65 | 59 | 67
  24-Hours: Excellent | 132 | 109 | 82 | 80

10. Secondary Outcome: Incidence and Type of Adverse Events
Description: The incidence of treatment emergent adverse events (TEAE) reported from first dose (Day 1) to last scheduled contact with the participant on Day 14 was descriptively summarized. Selected TEAEs were events with preferred terms of nausea, vomiting, abdominal pain, gastrointestinal bleeding, dizziness, or hypotension.
Time Frame: Day 1 to Day 14
Population: Safety Set
Measure: Number; unit: participants
Arm/Group | Tramadol/Diclofenac 50/50 | Tramadol/Diclofenac 25/25 | Tramadol 50 | Diclofenac 50
Number analyzed (Participants) | 208 | 205 | 206 | 207
participants
  TEAE | 96 | 62 | 105 | 48
  Severe TEAE | 6 | 1 | 3 | 2
  TEAE related to IMP or rescue medication | 49 | 23 | 64 | 10
  Serious TEAE | 0 | 1 | 0 | 0
  TEAE with outcome of death | 0 | 0 | 0 | 0
  Selected TEAE | 68 | 26 | 77 | 13
  TEAE leading to dose reduction | 0 | 0 | 0 | 0
  TEAE leading to dose interruption | 1 | 2 | 1 | 0
  TEAE leading to IMP withdrawal | 2 | 1 | 1 | 0
  Dose reduction, interruption, or withdrawal | 3 | 3 | 2 | 0

ADVERSE EVENTS:
Time Frame: Day 1 to Day 14
Description: Sites were instructed not to report dental pain as an AE until 24 hours after the first dose of IMP.
Arm/Group | Tramadol/Diclofenac 50/50 | Tramadol/Diclofenac 25/25 | Tramadol 50 | Diclofenac 50
All-Cause Mortality (participants affected / at risk) | 0/208 | 0/205 | 0/206 | 0/207
Serious Adverse Events (participants affected / at risk) | 0/208 | 1/205 | 0/206 | 0/207
Other Adverse Events (participants affected / at risk) | 96/208 | 62/205 | 105/206 | 48/207
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tramadol/Diclofenac 50/50 (N=208) | Tramadol/Diclofenac 25/25 (N=205) | Tramadol 50 (N=206) | Diclofenac 50 (N=207)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tramadol/Diclofenac 50/50 (N=208) | Tramadol/Diclofenac 25/25 (N=205) | Tramadol 50 (N=206) | Diclofenac 50 (N=207)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 51 (59) | 15 (17) | 52 (62) | 7 (7)
Oral pain (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 41 (57) | 12 (15) | 44 (75) | 3 (3)
Chills (General disorders) | 1 (1) | 3 (3) | 3 (3) | 1 (1)
Face oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inflammation (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 4 (4) | 6 (6) | 0 (0)
Alveolar osteitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Post procedural inflammation (Injury, poisoning and procedural complications) | 2 (2) | 4 (4) | 5 (5) | 3 (3)
Post procedural swelling (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 26 (26) | 21 (21) | 24 (24) | 18 (18)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 25 (28) | 11 (11) | 29 (34) | 6 (6)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 10 (10) | 6 (6) | 15 (16) | 7 (7)
Hypoaesthesia (Nervous system disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (6) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 2 (3) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor reserves the right to review any proposed presentation of the results of this trial before they are submitted for publication or public disclosure. Neither party (e.g., the sponsor, the coordinating investigator) has the right to prohibit publication or public disclosure unless it can be shown to affect possible patent rights.

DOCUMENTS (2):
  • Study Protocol (2017-10-19): https://cdn.clinicaltrials.gov/large-docs/72/NCT03714672/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-19): https://cdn.clinicaltrials.gov/large-docs/72/NCT03714672/SAP_001.pdf